CLINICAL TRIAL: NCT03064438
Title: A RANDOMIZED, DOUBLE-BLIND, VEHICLE CONTROLLED, PROOF-OF CONCEPT STUDY OF THE SAFETY AND EFFICACY OF ACU-D1 OINTMENT IN SUBJECTS WITH ACNE ROSACEA
Brief Title: Safety and Efficacy of ACU-D1 in the Treatment of Acne Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accuitis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACU-D1
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Acne Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACU-D1 Ointment (Experimental): Twice-daily application of ACU-D1 ointment to the face for 12 weeks.
  Interventions: Drug: ACCU-D1
- ACU-D1 Ointment Vehicle (Placebo Comparator): Twice-daily application of ACU-D1 ointment vehicle to the face for 12 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ACCU-D1 — ACCU-D1
  Arms: ACU-D1 Ointment
Drug: Vehicle — Placebo Comparator
  Arms: ACU-D1 Ointment Vehicle

SUMMARY:
The study evaluated the safety, tolerability, and efficacy of ACCU-D1 when applied twice daily for 12 weeks in adult participants with moderate to severe acne rosacea. Two-third of the participants received ACCU-D1 while one-third of the participants received vehicle control.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or non-pregnant and non-lactating female at least 18 years of age
* Participant has a clinical diagnosis of stable papulopustular rosacea (type-2)
* Participant has a total of ≥10 and ≤40 inflammatory lesions (papules, pustules, and nodules) on the face
* Participant has ≤2 nodules on the face
* Participant has an investigator's global assessment (IGA) score of ≥3
* If the participant is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an approved effective method of birth control for the duration of the study
* Participant is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of rosacea or which exposes the participant to an unacceptable risk by study participation
* Participant is willing and able to follow all study instructions and to attend all study visits
* Participant is able to comprehend and willing to sign an informed consent form

Exclusion Criteria:

* Participant is pregnant, nursing, or planning to become pregnant during the duration of the study
* Participant has used systemic glucocorticosteroids within 42 days prior to Visit 1 (inhaled and ocular glucocorticosteroids are permitted)
* Participant has used systemic antibiotics within 28 days prior to Visit 1
* Participant has used any topical glucocorticosteroids on the face within 28 days prior to Visit 1
* Participant has used any prescription or over-the-counter product for the treatment of acne or rosacea within 14 days prior to Visit 1
* Participant is currently using any therapy that, in the investigator's opinion, is a photosensitizer (for example, phenothiazines, amiodarone, quinine, thiazides, sulphonamides, quinolones, etc.)
* Participant currently has any skin disease (for example, psoriasis, atopic dermatitis, eczema), or condition (for example, actinic keratosis, photo-damage, sunburn, excessive hair, open wounds) that, in the investigator's opinion, might impair evaluation of rosacea or which exposes the subject to an unacceptable risk by study participation
* Participant currently has, on the face, or has had on the face, any of the following within the specified period prior to Visit 1 that, in the investigator's opinion, might impair evaluation of rosacea or which exposes the subject to an unacceptable risk by study participation:

  * A cutaneous malignancy; 180 days
  * Experienced a sunburn; 14 days
* Participant has facial hair, that in the investigator's opinion, might impair evaluation of rosacea or proper study medication application
* Participant has a history of sensitivity to any of the ingredients in the study medications
* Participant has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DS Research, Louisville, Kentucky
  - DermResearch, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson JM, Coulon R, Arbiser JL. Evaluation of a First-in-Class Proteasome Inhibitor in Patients With Moderate to Severe Rosacea. J Drugs Dermatol. 2021 Jun 1;20(6):660-664. doi: 10.36849/JDD.2021.5925. PMID 34076401

FDAAA 801 VIOLATIONS:
- Correction Confirmed — The responsible party has corrected the violation. — issued 2022-05-26, released 2021-08-17, posted 2022-06-07
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2021-07-26, released 2018-04-12, posted 2021-07-29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two sites in the United States.
Pre-assignment Details: Eligible participants will be assigned in a random manner to 1 of the 2 study medications in a 2:1 ratio (ACU-D1 ointment: ACU-D1 ointment vehicle).
Period: Overall Study
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Started | 27 | 13
Completed | 26 | 12
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (MITT) population included all randomized participants who were dispensed study medication and provided any post-baseline efficacy data.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle | Total
Number analyzed (Participants) | 27 | 13 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.59 (11.537) | 51.08 (12.473) | 50.08 (11.708)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 22 | 13 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 13 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total lesion count [Mean (Standard Deviation); unit: number of lesions] — Total lesion count was the sum of counts of the following lesion types (face only): Papule - raised inflammatory lesions, < 0.5 cm in diameter with no visible purulent material; Pustule - raised inflammatory lesions, < 0.5 cm in diameter with visible purulent material; Nodule - any circumscribed, inflammatory mass ≥ 0.5 cm in diameter.
  number of lesions | 18.00 (9.413) | 20.46 (9.777) | 18.80 (9.479)
Erythema score based on local tolerability as assessed by the investigator [Count of Participants; unit: Participants] — Erythema score at baseline (pre-application) was evaluated by the investigator on a 0 to 3 scale with a lower score indicating lesser severity.
  Score 0 (clear): no erythema present; Score 1 (mild): slight erythema; Score 2 (moderate): definite erythema; Score 3 (severe): marked, fiery erythema. The assessment was based on the safety population which included all randomized participants who received at least 1 dose of study medication.
  Participants
    Score 0 (clear) | 1 | 1 | 2
    Score 1 (mild) | 5 | 4 | 9
    Score 2 (moderate) | 16 | 5 | 21
    Score 3 (severe) | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Lesion Count at Week 12
Description: Total lesion count was the sum of counts of the following lesion types (face only): Papule - raised inflammatory lesions, <0.5 cm in diameter with no visible purulent material; Pustule - raised inflammatory lesions, <0.5 cm in diameter with visible purulent material; Nodule - any circumscribed, inflammatory mass ≥0.5 cm in diameter.
Time Frame: Baseline, Week 12
Population: Number of participants included participants in the MITT population with available data at Week 12.
Measure: Least Squares Mean (Standard Error); unit: number of lesions
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 26 | 11
number of lesions | -10.2 (1.08) | -12.0 (1.62)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Test type: Superiority; p = 0.366, t-test, 2 sided; Difference of Least Squares (LS) Mean = 1.8, 95% CI 2-sided [-2.162 to 5.727], Standard Error of Mean 1.95

2. Secondary Outcome: Percent Change From Baseline in Investigator's Global Assessment (IGA) Score at Weeks 2, 4, 8, and 12
Description: The IGA score is an ordered categorical value ranging from 0 (clear) to 4 (severe). A lower score indicated improvement in the condition.
  Score 0 (clear): no papules or pustules, no nodules, none or barely perceptible erythema
  Score 1 (near clear): very few (≤3) papules and/or pustules, no nodules, very mild erythema
  Score 2 (mild): few papules and pustules present, no nodules, mild erythema
  Score 3 (moderate): several papules and pustules are the predominant features, ≤2 nodules may be present, moderate erythema
  Score 4 (severe): numerous papules and pustules, multiple nodules may be present, severe erythema
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: MITT population. Number of participants analyzed included participants with available data at specific timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
percent change
  Week 2 | -23 (0.2561) | -29 (0.1653)
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4 | -35 (0.2387) | -26 (0.2771)
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8 | -31 (0.2538) | -29 (0.2233)
  Week 12: number analyzed (Participants) | 26 | 11
  Week 12 | -31 (0.2588) | -26 (0.3583)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Percent change from baseline at Week 2; Test type: Superiority; p = 0.1099, Van Elteren test
Statistical Analysis 2: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Percent change from baseline at Week 4; Test type: Superiority; p = 0.1653, Van Elteren test
Statistical Analysis 3: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Percent change from baseline at Week 8; Test type: Superiority; p = 0.8437, Van Elteren test
Statistical Analysis 4: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Percent change from baseline at Week 12; Test type: Superiority; p = 0.4644, Van Elteren test

3. Secondary Outcome: Percentage of Participants Who Were Treatment Responders at Week 12
Description: Treatment responders were defined as participants who have either (1) 2 ordinal or more reductions in the IGA score from baseline or (2) an IGA score of 0 or 1.
  The IGA score is an ordered categorical value ranging from 0 (clear) to 4 (severe). A lower score indicated improvement in the condition.
  Score 0 (clear): no papules or pustules, no nodules, none or barely perceptible erythema
  Score 1 (near clear): very few (≤3) papules and/or pustules, no nodules, very mild erythema
  Score 2 (mild): few papules and pustules present, no nodules, mild erythema
  Score 3 (moderate): several papules and pustules are the predominant features, ≤2 nodules may be present, moderate erythema
  Score 4 (severe): numerous papules and pustules, multiple nodules may be present, severe erythema
Time Frame: Baseline, Week 12
Population: MITT population. Number of participants analyzed included participants with available IGA score at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 26 | 11
percentage of participants | 19.2 | 18.2
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Test type: Superiority; p = 1.0, Fisher Exact

4. Secondary Outcome: Change From Baseline in Papule Lesions at Weeks 2, 4, 8, and 12
Description: Papule - raised inflammatory lesions, <0.5 cm in diameter with no visible purulent material
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: MITT population. Number of participants analyzed included participants with available data at specified visits.
Measure: Least Squares Mean (Standard Error); unit: number of lesions
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
number of lesions
  Week 2 | -6.6 (1.09) | -7.95 (1.57)
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4 | -9.7 (0.97) | -8.22 (1.44)
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8 | -8.1 (1.16) | -10.30 (1.71)
  Week 12: number analyzed (Participants) | 26 | 11
  Week 12 | -9.2 (1.01) | -10.98 (1.53)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 2; Test type: Superiority; p = 0.495, t-test, 2 sided; Difference of LS Mean = 1.3, 95% CI 2-sided [-2.571 to 5.211], Standard Error of Mean 1.91
Statistical Analysis 2: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 4; Test type: Superiority; p = 0.399, t-test, 2 sided; Difference of LS Mean = -1.5, 95% CI 2-sided [-5.014 to 2.045], Standard Error of Mean 1.74
Statistical Analysis 3: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 8; Test type: Superiority; p = 0.290, t-test, 2 sided; Difference of LS Mean = 2.2, 95% CI 2-sided [-1.965 to 6.407], Standard Error of Mean 2.07
Statistical Analysis 4: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 12; Test type: Superiority; p = 0.343, t-test, 2 sided; Difference of LS Mean = 1.8, 95% CI 2-sided [-1.953 to 5.469], Standard Error of Mean 1.83

5. Secondary Outcome: Change From Baseline in Pustule Lesions at Weeks 2, 4, 8, and 12
Description: Pustule - raised inflammatory lesions, <0.5 cm in diameter with visible purulent material
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: MITT population. Number of participants analyzed included participants with available data at specified visits.
Measure: Least Squares Mean (Standard Error); unit: number of lesions
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
number of lesions
  Week 2 | -0.4 (0.43) | -0.98 (0.62)
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4 | -1.2 (0.20) | -1.63 (0.30)
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8 | -1.1 (0.25) | -1.29 (0.38)
  Week 12: number analyzed (Participants) | 26 | 11
  Week 12 | -1.0 (0.31) | -1.04 (0.48)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 2; Test type: Superiority; p = 0.407, t-test, 2 sided; Difference of LS Mean = 0.6, 95% CI 2-sided [-0.894 to 2.155], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 4; Test type: Superiority; p = 0.291, t-test, 2 sided; Difference of LS Mean = 0.4, 95% CI 2-sided [-0.342 to 1.109], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 8; Test type: Superiority; p = 0.734, t-test, 2 sided; Difference of LS Mean = 0.2, 95% CI 2-sided [-0.763 to 1.073], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline in pustule lesions at Week 12; Test type: Superiority; p = 0.952, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-1.128 to 1.197], Standard Error of Mean 0.57

6. Secondary Outcome: Change From Baseline in Nodule Lesions at Weeks 2, 4, 8, and 12
Description: Nodule - any circumscribed, inflammatory mass ≥0.5 cm in diameter
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: MITT population. Number of participants analyzed included participants with available data at specified visits.
Measure: Least Squares Mean (Standard Error); unit: number of lesions
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
number of lesions
  Week 2 | 0.0 (0.04) | 0.02 (0.06)
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4 | 0.0 (0.04) | -0.05 (0.06)
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8 | 0.0 (0.04) | -0.05 (0.06)
  Week 12: number analyzed (Participants) | 26 | 11
  Week 12 | 0.0 (0.04) | 0.04 (0.06)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 2; Test type: Superiority; p = 0.313, t-test, 2 sided; Difference of LS Mean = -0.1, 95% CI 2-sided [-0.215 to 0.069], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 4; Test type: Superiority; p = 0.942, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.141 to 0.152], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline in nodule lesions at Week 8; Test type: Superiority; p = 0.284, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [-0.067 to 0.226], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 12; Test type: Superiority; p = 0.542, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.198 to 0.105], Standard Error of Mean 0.08

7. Secondary Outcome: Change From Baseline in Papules + Pustules Lesions at Weeks 2, 4, 8, and 12
Description: Papules + pustules lesions were the sum of counts of papule (raised inflammatory lesions, <0.5 cm in diameter with no visible purulent material) and pustule (raised inflammatory lesions, <0.5 cm in diameter with visible purulent material) lesions.
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: MITT population. Number of participants analyzed included participants with available data at specified visits.
Measure: Least Squares Mean (Standard Error); unit: number of lesions
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
number of lesions
  Week 2 | -7.0 (1.16) | -8.97 (1.67)
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4 | -10.9 (1.06) | -9.90 (1.57)
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8 | -9.2 (1.19) | -11.65 (1.75)
  Week 12: number analyzed (Participants) | 26 | 11
  Week 12 | -10.2 (1.08) | -12.03 (1.62)
Statistical Analysis 1: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 2; Test type: Superiority; p = 0.333, t-test, 2 sided; Difference of LS Mean = 2.0, 95% CI 2-sided [-2.135 to 6.139], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 4; Test type: Superiority; p = 0.591, t-test, 2 sided; Difference of LS Mean = -1.0, 95% CI 2-sided [-4.882 to 2.822], Standard Error of Mean 1.90
Statistical Analysis 3: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 8; Test type: Superiority; p = 0.254, t-test, 2 sided; Difference of LS Mean = 2.5, 95% CI 2-sided [-1.840 to 6.758], Standard Error of Mean 2.12
Statistical Analysis 4: Comparison: ACU-D1 Ointment vs ACU-D1 Ointment Vehicle; Change from baseline at Week 12; Test type: Superiority; p = 0.356, t-test, 2 sided; Difference of LS Mean = 1.8, 95% CI 2-sided [-2.131 to 5.779], Standard Error of Mean 1.95

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants reporting any adverse event including local tolerability of signs and symptoms of irritation, clinical laboratory safety tests, and vital signs.
Time Frame: Baseline to Week 14
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
Participants | 11 | 4

9. Other Pre Specified Outcome: Number of Participants With Erythema Score Based on Local Tolerability as Assessed by the Investigator at Week 12
Description: Erythema score was evaluated by the investigator on a 0 to 3 scale with a lower score indicating lesser severity.
  Score 0 (clear): no erythema present
  Score 1 (mild): slight erythema
  Score 2 (moderate): definite erythema
  Score 3 (severe): marked, fiery erythema
Time Frame: Week 12
Population: Safety population included all randomized participants who received at least 1 dose of study medication. Number of participants analyzed included participants with available data at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 26 | 11
Participants
  Score 0 (clear) | 1 | 1
  Score 1 (mild) | 14 | 3
  Score 2 (moderate) | 9 | 6
  Score 3 (severe) | 2 | 1

10. Other Pre Specified Outcome: Number of Participants With Erythema Score Based on Local Tolerability as Assessed by the Investigator at Day 1 (Post-application) and Weeks 2, 4, 8, and 14
Description: as for outcome 9
Time Frame: Day 1 (Post-application) and Weeks 2, 4, 8, and 14
Population: Safety population. Number of participants analyzed included participants with available data at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
Number analyzed (Participants) | 27 | 13
Participants
  Day 1 (Post-application): Score 0 (clear) | 1 | 1
  Day 1 (Post-application): Score 1 (mild) | 9 | 4
  Day 1 (Post-application): Score 2 (moderate) | 12 | 4
  Day 1 (Post-application): Score 3 (severe) | 5 | 4
  Week 2: Score 0 (clear) | 0 | 0
  Week 2: Score 1 (mild) | 12 | 7
  Week 2: Score 2 (moderate) | 12 | 4
  Week 2: Score 3 (severe) | 3 | 2
  Week 4: number analyzed (Participants) | 27 | 12
  Week 4: Score 0 (clear) | 0 | 0
  Week 4: Score 1 (mild) | 13 | 4
  Week 4: Score 2 (moderate) | 12 | 7
  Week 4: Score 3 (severe) | 2 | 1
  Week 8: number analyzed (Participants) | 27 | 12
  Week 8: Score 0 (clear) | 1 | 1
  Week 8: Score 1 (mild) | 11 | 5
  Week 8: Score 2 (moderate) | 13 | 6
  Week 8: Score 3 (severe) | 2 | 0
  Week 14: number analyzed (Participants) | 26 | 12
  Week 14: Score 0 (clear) | 2 | 1
  Week 14: Score 1 (mild) | 8 | 3
  Week 14: Score 2 (moderate) | 13 | 5
  Week 14: Score 3 (severe) | 3 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 14
Description: Safety population
Arm/Group | ACU-D1 Ointment | ACU-D1 Ointment Vehicle
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 11/27 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACU-D1 Ointment (N=27) | ACU-D1 Ointment Vehicle (N=13)
Vomiting (Gastrointestinal disorders) | 1 | 0
Administration site dryness (General disorders) | 1 | 1
Administration site warmth (General disorders) | 1 | 0
Application site perspiration (General disorders) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03064438/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03064438/SAP_001.pdf